CLINICAL TRIAL: NCT03929783
Title: Improving PPV3 Using Contrast Enhanced Mammography (CEM) in Diagnostic Assessment by Reducing Benign Tissue Diagnosis (FP3) - A Single-Arm Prospective Study
Brief Title: Contrast Enhanced Mammography in Diagnosing Patients With Suspicious Breast Findings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19D.203; JT 13786 (Other: JeffTrial Number)
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (CEM) (Experimental): Patients undergo contrast enhanced mammography prior to scheduled standard of care core needle biopsy of the breast on the same day.
  Interventions: Procedure: Contrast Enhanced Digital Mammography

INTERVENTIONS:
Procedure: Contrast Enhanced Digital Mammography — Undergo CEM
  Other Names: CEDM; Contrast Enhanced Spectral Mammography

SUMMARY:
This pilot trial studies how well contrast enhanced mammography works in diagnosing patients with suspicious breast findings. Diagnostic procedures, such as contrast enhanced mammography, may help to reclassify findings seen on diagnostic mammography and ultrasound as benign or likely benign with what would otherwise require biopsy for confirmation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary data to support the hypothesis that contrast enhanced mammography (CEM) can reduce benign tissue diagnosis (FP3) and therefore improve positive predictive value 3 (PPV3).

SECONDARY OBJECTIVES:

I. Identify specific CEM characteristics that accurately classify a finding as benign, high-risk or malignant.

II. Assess the positive and negative predictive values for each digital breast tomosynthesis (DBT), breast ultrasound and CEM.

EXPLORATORY OBJECTIVES:

I. To compare the outcomes/endpoints stratified by age to determine if age affects the ability of CEM to accurately define a lesion as benign, probably benign or suspicious.

OUTLINE:

Patients undergo contrast enhanced mammography prior to scheduled standard of care core needle biopsy of the breast on the same day or up to 3 days later.

ELIGIBILITY:
Inclusion Criteria:

* Women with digital breast tomosynthesis and/or ultrasound assessments of Breast Imaging Reporting and Data System (BI-RADS) 4 and 5 lesions with recommendation of needle biopsy for tissue diagnosis.
* Abnormal findings include masses, focal, global or developing asymmetries, architecture distortions, or > 1 cm of suspicious calcifications with or without associated ultrasound abnormal findings.
* Scheduled for imaging guided percutaneous needle biopsy.
* Provide signed and dated informed consent form.
* If patient is of childbearing potential, a negative pregnancy test, urine or blood, within 14 days prior to the scan.

Exclusion Criteria:

* < 1 cm span of calcifications without an ultrasound correlate.
* Pregnant patients.
* Patients with known allergy to iodinated contrast material.
* If patient answers YES to any of the below questions they need glomerular filtration rate (gFR) prior to contrast administration regardless of their age:

  * Have you ever been told you have renal problems?
  * Have you ever been told you have protein in your urine?
  * Do you have high blood pressure?
  * Do you have diabetes?
  * Do you have gout?
  * Have you ever had kidney surgery?

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Sensitivity of contrast enhanced mammography (CEM) to classify a lesion as benign, probably benign, or suspicious | Up to 1 year
  The total number of suspicious and benign lesions on each modality (mammogram+ultrasound [MM+US] and CEM) will be calculated and compared to a final tissue diagnosis independently.
Sensitivity of MM to classify a lesion as benign, probably benign, or suspicious | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
Sensitivity of US to classify a lesion as benign, probably benign, or suspicious | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
Specificity of CEM to classify a lesion as benign, probably benign, or suspicious | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
Specificity of MM to classify a lesion as benign, probably benign, or suspicious | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
Specificity of US to classify a lesion as benign, probably benign, or suspicious | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
False negative rate of CEM | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
False negative rate of MM | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
False negative rate of US | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
False positive rate of CEM | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
False positive rate of MM | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.
False positive rate of US | Up to 1 year
  The total number of suspicious and benign lesions on each modality (MM+US and CEM) will be calculated and compared to a final tissue diagnosis independently.

SECONDARY OUTCOMES:
Positive predictive value of CEM | Up to 1 year
  The positive predictive value of CEM will be calculated and compared to MM+US.
Positive predictive value of MM | Up to 1 year
  The positive predictive value of CEM will be calculated and compared to MM+US.
Positive predictive value of US | Up to 1 year
  The positive predictive value of CEM will be calculated and compared to MM+US.
Negative predictive value of CEM | Up to 1 year
  The negative predictive value of CEM will be calculated and compared to MM+US.
Negative predictive value of MM | Up to 1 year
  The negative predictive value of CEM will be calculated and compared to MM+US.
Negative predictive value of US | Up to 1 year
  The negative predictive value of CEM will be calculated and compared to MM+US.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Liao, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States